## STUDY PROTOCOL

Storage symptoms are experienced during the storage phase of the bladder and include daytime frequency and nocturia. The Standardization Committee of the International Continence Society (ICS) defined increased bladder sensation as "symptoms such as feeling of an early and persistent desire to void".

The aim of this study is to assess the effectiveness of medium frequency electrotherapy (interferential currents) treatment for increased bladder sensation, urgency and LUTS.

Design: Quasi-experimental, longitudinal, pre-/post-. Level of evidence II/III. Case-control study, non-randomized inclusion of consecutive type.

Informed consent before inclusion in the study, as established by the Declaration of Helsinki.

Statistical analysis of data using SPSS 22.0 for Windows.

Statistical methods: descriptive statistics for quantitative variables (procedure DESCRIPTIVE) and descriptive statistics for qualitative variables (FREQUENCIES procedure), contingency tables for the relationship between qualitative variables (procedure CROSSTABS, chi-square test and T-student). A p<0.005 is considered significant.

| Cases vs Controls | |
|-------------------|----------------------------------------------------------|
| P01 | Age (years) |
| P02 | Age |
| P03 | Age of UI symptom |
| P04 | Urinary incontinence |
| P05 | Urgency |
| P06 | Increased daytime frequency |
| P07 | Nocturia |
| P08 | Nocturnal enuresis |
| P09 | Pelvic pain |
| P10 | Feeling of prolapse |
| P11 | UTI |
| P12 | Constipation |
| P13 | Feeling incomplete emptying |
| P14 | Burning urination |
| P15 | Lower urinary tract symptoms |
| P16 | Overactive bladder |
| P17 | Urinary stress incontinence |
| P18 | Urgency feeling |
| P19 | Bladder outlet obstruction |
| P20 | Urine flow |
| P21 | Sessions of treatment |
| P22 | Discharge / End of treatment due to clinical improvement |
| P23 | Urinary incontinence post- |
| P24 | Urgency post- |
| P25 | Increased daytime frequency post- |
| P26 | Nocturia post- |
| P27 | Nocturnal enuresis post- |
| P28 | Pelvic pain post- |
| P29 | Feeling incomplete emptying post- |
| P30 | Burning urination post- |
| P31 | Lower urinary tract symptoms post- |